CLINICAL TRIAL: NCT07199829
Title: A Double-Blind Randomized Controlled Trial Evaluating Response to Vitamin D3 and K2 Supplementation Through Inflammatory Markers and the Gut Microbiome in Healthcare Personnel
Brief Title: Evaluating Response to Vitamin D3 and K2 Supplementation in Healthcare Personnel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary S McCarthy, Senior Nurse Scientist, Madigan Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 225015; 11207-N24-B11 (Other Grant/Funding Number: TriService Nursing Research Program / USUHS)
Record Dates: First submitted 2025-02-06; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hypovitaminosis D; Hypovitaminosis
Keywords: Hypovitaminosis D; Hypovitaminosis K; Gut microbiome
MeSH Terms: conditions — Vitamin D Deficiency; Avitaminosis

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial (RCT) with 4 arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin Arm 1 (Active Comparator): Vitamin D3 125 mcg taken orally once daily for 90 days
  Interventions: Dietary Supplement: Vitamin Arm 1
- Vitamin Arm 2 (Active Comparator): Vitamin K2 180 mcg taken orally once daily for 90 days
  Interventions: Dietary Supplement: Vitamin Arm 2
- Vitamin Arm 3 (Active Comparator): Vitamin D3 125 mcg combined with vitamin K2 180 mcg taken orally once daily for 90 days
  Interventions: Dietary Supplement: Vitamin Arm 3
- Placebo Arm (Placebo Comparator): Inert capsule taken orally once daily for 90 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin Arm 1 — Subject receives dietary supplement for 90 days
  Arms: Vitamin Arm 1
Dietary Supplement: Vitamin Arm 2 — Subject receives dietary supplement for 90 days
  Arms: Vitamin Arm 2
Dietary Supplement: Vitamin Arm 3 — Subject receives dietary supplement for 90 days
  Arms: Vitamin Arm 3
Other: Placebo — Subject receives placebo for 90 days
  Arms: Placebo Arm

SUMMARY:
The main purpose of this research study is to learn about the effects of supplemental vitamin D3 and vitamin K2 on blood levels and the gut microbial community, called the gut microbiome. There are many influences on blood levels of vitamin D and K to include your dietary intake, lifestyle behaviors (physical activity, sleep), genetic alterations in metabolism of these vitamins, and the gut microbial abundance and diversity. You will be asked to take one capsule containing vitamin D3 (125 mcg), vitamin K2 (180 mcg), a combination of vitamins D3 and K2 (same doses as previous), or a placebo powder for 90 days. You will also be asked to complete questionnaires, undergo body composition and blood pressure measurements, provide blood samples and a stool swab, all on 2 occasions about 3 - 4 months apart. By conducting this study, we aim to identify the frequency of common genetic alterations in vitamins D and K metabolism and establish the impact on the gut microbiome for the first time. Your participation in this study will last about 4 - 6 months and include up to 3 visits.

DETAILED DESCRIPTION:
Health promotion efforts for all branches of Service aim to ensure the health and readiness of the Force. This timely, relevant study supports this effort as well as the TriService Nursing Research Program priorities of Fit and Ready Force, Care for the Caregiver, and Translate Research into Practice. In 2023, the Defense Health Agency unveiled its strategic plan through 2028 which included these two priorities, 1) 'achieving new levels of excellence by fully leveraging emerging scientific and technological advancements to optimize the health and care experience of our beneficiaries', and 2) 'creating a workplace where people are the primary focus, and the principles of high reliability nurture and energize each individual'. The previous nutrigenomics work by this research team, the expertise and enthusiasm of our new members, and the choice of diverse cohorts for this study, presents an exciting and potentially impactful extension of nutrigenomics with metagenomics of the gut microbiome to provide insight into complex nutrient pathways and specifically, the response of the gut microbial community to select micronutrients. Vitamin D and vitamin K2 are vital micronutrients that support immune, bone, gut, and cardiometabolic health with insufficiencies contributing to musculoskeletal injuries (MSKi), metabolic syndrome, cardiovascular disease, and gut dysbiosis. This Follow-On research application advances the science linking vitamin D, lifestyle behaviors, and chronic disease prevention in healthy adults by probing unexplored areas such as a key symbiotic nutrient, vitamin K2, with vitamin D3, next generation sequencing (NGS) of polymorphisms involved in vitamin metabolism pathways as well as metagenomics to assess the response of the gut microbial community to dietary and supplemental nutrients. The Specific Aims and research questions for our study include:

Specific Aim 1. Evaluate effect of vitamin D3 and K2 dietary intake and supplementation groups vs placebo group on the gut microbiome; Research Question (RQ)1.a. Will gut microbiome composition, diversity, and richness respond differently to each treatment group - vitamin D3, vitamin K2, D3+K2 versus the control group? RQ1.b. What effect will vitamin D3 and/or K2 metabolism pathway single nucleotide polymorphisms (SNPs) have on gut microbiome response?

Specific Aim 2. Assess response to vitamin supplementation with serum 25-hydroxyvitamin D [25(OH)D] and osteocalcin levels pre and post supplement; RQ2. Will selected doses, based on clinical experience and published data, achieve designated endpoints for sufficiency; serum 25(OH)D greater than 30 ng/mL and undercarboxylated osteocalcin (ucOC) within normal limits?

Specific Aim 3. Assess the influence of vitamin D and K metabolism pathway SNPs on serum 25(OH)D and osteocalcin to determine vitamin D3, K2, and D3 + K2 supplementation efficacy; RQ3. To what extent does the presence of vitamin D and/or K metabolism pathway SNPs affect supplement efficacy when comparing treatment vs control group response measured by serum biomarkers?

Specific Aim 4. Explore relationships between diet/Dietary Inflammatory Index (DII), lifestyle behaviors (steps and sleep), body composition, metabolic and inflammatory biomarkers, SNPs, and the gut microbiome from Baseline to 3 months; RQ4.a. What factors need consideration when exploring genetic and non-genetic contributions to the gut microbiome in the treatment vs control group? RQ4.b. What role do age, gender, body mass index, inflammation status, and lipid profile play in the gut microbiome composition?

Hypothesis 1: Genotypic alterations in vitamin D3 and/or K2 metabolism pathways will influence gut microbiome composition in response to supplementation.

Hypothesis 2: Genotypic alterations in vitamin D3 and/or K2 metabolism pathways will influence serum response to supplementation.

ELIGIBILITY:
Inclusion Criteria:

* able to read and understand English
* 25 OHD serum level equal to or less than 30 ng/mL
* willing to discontinue vitamin D3 and/or K2 supplements for 4.5 months
* military beneficiary (Active Duty, Retired, Dependent)
* remaining employed at workplace for 6 months

Exclusion Criteria:

* Diagnosed medical condition that prevents nutrient absorption from food (e.g. Inflammatory Bowel Disease, Celiac Disease, post-Roux-en-Y/Gastric sleeve surgery)
* Pregnant or breastfeeding
* Current antibiotic use or within past 3 months
* Current anticoagulant use or within past 3 months
* Current weight loss or fat malabsorption medication use (e.g. Glucagon-Like Peptide 1 agonists, Orlistat)
* Allergies or sensitivities to methylcellulose, vitamin D (D3, D2), or vitamin K (K2, Menaquinone-4, Menaquinone-7)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome composition | 90 days
  Evaluate effect of vitamin D3 and K2 dietary intake, and assigned vitamin supplementation group versus placebo group, on the gut microbiome composition
Gut microbiome richness | 90 days
  Will use Operational Taxonomic Units, Simpson Index and /or Chao1 index to evaluate gut microbiome richness before and after vitamin supplementation vs placebo
Gut microbiome diversity | 90 days
  Will use Operational Taxonomic Units, Simpson Index and /or Chao1 index to evaluate gut microbiome diversity before and after vitamin supplementation vs placebo

SECONDARY OUTCOMES:
Serum 25OHD | 90 days
  Response to vitamin supplementation with serum 25(OH)D level pre and post supplement
Serum Osteocalcin level | 90 days
  Response to vitamin supplementation with serum osteocalcin level pre and post supplement
Vitamin D3 and K2 metabolic pathway variants on supplementation efficacy | 90 days
  Examine vitamin D3 and K2 metabolism pathway single nucleotide polymorphisms for effect on serum 25(OH)D and osteocalcin levels
Genetic and non-genetic factor contributions to gut microbiome composition | 90 days
  Explore relationships between diet, lifestyle behaviors (steps and sleep), body composition, metabolic and inflammatory serum biomarkers, and single nucleotide polymorphisms, and the gut microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Mary S McCarthy, PhD, Principal Investigator — Madigan AMC
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A data sharing agreement has been developed and submitted to the Defense Health Agency; approval has been received.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Supporting information will be available upon request after completion of protocol, for the following 2 years.
Access Criteria: Contact principal investigator at mary.s.mccarthy1.civ@health.mil

REFERENCES:
- [Background] Akimbekov NS, Digel I, Sherelkhan DK, Lutfor AB, Razzaque MS. Vitamin D and the Host-Gut Microbiome: A Brief Overview. Acta Histochem Cytochem. 2020 Jun 26;53(3):33-42. doi: 10.1267/ahc.20011. Epub 2020 Jun 16. PMID 32624628
- [Background] Levin GP, Robinson-Cohen C, de Boer IH, Houston DK, Lohman K, Liu Y, Kritchevsky SB, Cauley JA, Tanaka T, Ferrucci L, Bandinelli S, Patel KV, Hagstrom E, Michaelsson K, Melhus H, Wang T, Wolf M, Psaty BM, Siscovick D, Kestenbaum B. Genetic variants and associations of 25-hydroxyvitamin D concentrations with major clinical outcomes. JAMA. 2012 Nov 14;308(18):1898-905. doi: 10.1001/jama.2012.17304. PMID 23150009
- [Background] Ammar M, Heni S, Tira MS, Khalij Y, Hamdouni H, Amor D, Ksibi S, Omezzine A, Bouslama A. Variability in response to vitamin D supplementation according to vitamin D metabolism related gene polymorphisms in healthy adults. Eur J Clin Nutr. 2023 Feb;77(2):189-194. doi: 10.1038/s41430-022-01218-y. Epub 2022 Sep 27. PMID 36167979